CLINICAL TRIAL: NCT07403994
Title: The Longitudinal Impact of Prenatal Pilates on Female Sexual Function and Sexual Distress During Pregnancy
Brief Title: Prenatal Pilates and Sexual Function During Pregnancy
Acronym: PP-SEX
Status: Recruiting | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Gökçenur Karakelleoğlu, Assistant Professor of Obstetrics and Gynecology, Okan University
Other Study IDs: OKAN-PP-FSFI-2025
Record Dates: First submitted 2026-01-28; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Female Sexual Function During Pregnancy; Pregnancy; Female Sexual Function
Keywords: Pregnancy; Prenatal Pilates; Female Sexual Function; Sexual Distress; FSFI; FSDS-R; Physical Activity; Quality of Life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prenatal Pilates Group: Pregnant women who regularly participate in instructor-led prenatal Pilates during pregnancy by personal choice. Pilates sessions are performed in external Pilates studios under the supervision of certified instructors. No exercise program is prescribed, modified, or supervised by the study investigators. Participation in Pilates reflects usual lifestyle behavior.
- Control Group: Pregnant women who do not participate in prenatal Pilates or any structured exercise program during pregnancy and continue their usual daily activities without engaging in organized physical exercise.

SUMMARY:
Pregnancy is a period associated with significant hormonal, physical, and emotional changes that may affect a woman's sexual function and increase sexual distress. Sexual dysfunction and related distress are common during pregnancy and may negatively impact quality of life and intimate relationships.

Regular physical activity during pregnancy has been shown to improve physical well-being, emotional health, and overall quality of life. Prenatal Pilates is a commonly preferred exercise method among pregnant women and is thought to improve posture, pelvic floor muscle strength, body awareness, and stress levels. However, limited evidence exists regarding the effects of prenatal Pilates on female sexual function and sexual distress during pregnancy.

This prospective observational cohort study aims to evaluate changes in female sexual function and sexual distress throughout pregnancy and to compare these changes between pregnant women who regularly participate in instructor-led prenatal Pilates and those who do not engage in structured exercise. Participants will be enrolled during the first trimester and followed across all three trimesters of pregnancy.

Female sexual function will be assessed using the Female Sexual Function Index (FSFI), and sexual distress will be measured using the Female Sexual Distress Scale-Revised (FSDS-R). These questionnaires will be administered online during the first, second, and third trimesters. The study does not involve any intervention or exercise prescription; participants in the Pilates group will continue their usual prenatal Pilates activities by personal choice.

The results of this study are expected to contribute to a better understanding of the relationship between prenatal physical activity and sexual health during pregnancy and may help inform future counseling and supportive care strategies for pregnant women.

DETAILED DESCRIPTION:
Pregnancy is accompanied by substantial physiological, hormonal, and psychosocial changes that may influence female sexual function and contribute to increased sexual distress. Alterations in body image, fatigue, hormonal fluctuations, and emotional well-being during pregnancy have been associated with decreased sexual desire, arousal, and satisfaction. Despite the high prevalence of sexual dysfunction during pregnancy, this topic remains under-discussed in routine antenatal care.

Physical activity during pregnancy has been associated with multiple maternal benefits, including improved musculoskeletal function, reduced stress, and enhanced quality of life. Prenatal Pilates is a low-impact exercise modality that focuses on posture, breathing, pelvic floor muscle activation, core stabilization, and flexibility. It is commonly practiced by pregnant women and is considered safe when performed under the supervision of a certified instructor. While prenatal Pilates has been shown to improve physical comfort and psychological well-being, evidence regarding its association with female sexual function and sexual distress during pregnancy remains limited.

This study is designed as a prospective observational cohort study conducted at a single tertiary care center. Pregnant women with singleton pregnancies will be enrolled during the first trimester and followed longitudinally throughout pregnancy. Participants will be categorized into two groups based on their self-reported exercise behavior: those who regularly participate in instructor-led prenatal Pilates and those who do not engage in structured exercise during pregnancy. No exercise intervention or behavioral modification will be introduced as part of the study protocol.

Data will be collected using validated, self-administered questionnaires delivered through secure online platforms during the first, second, and third trimesters of pregnancy. Female sexual function will be assessed using the Female Sexual Function Index (FSFI), a 19-item instrument evaluating six domains of sexual function: desire, arousal, lubrication, orgasm, satisfaction, and pain. Sexual distress will be measured using the Female Sexual Distress Scale-Revised (FSDS-R), a 13-item questionnaire assessing sexually related personal distress. Higher FSFI scores indicate better sexual function, whereas higher FSDS-R scores reflect greater sexual distress.

Demographic and obstetric characteristics, including maternal age, parity, gestational age, and relevant medical history, will be collected at baseline. The primary objective of the study is to evaluate longitudinal changes in FSFI and FSDS-R scores across pregnancy. Secondary objectives include comparing temporal patterns of sexual function and distress between the prenatal Pilates and non-exercising groups.

Statistical analyses will be performed using appropriate longitudinal analytical methods. Within-group changes across trimesters will be assessed using repeated-measures analyses, while between-group differences over time will be evaluated using mixed-effects models or equivalent generalized linear modeling approaches, depending on data distribution. These analyses aim to account for both time-dependent changes and group-level differences.

This study seeks to provide further insight into the relationship between prenatal physical activity and sexual health during pregnancy. By examining sexual function and distress longitudinally, the findings may support more comprehensive counseling approaches and contribute to the growing body of evidence regarding non-pharmacological strategies to support sexual well-being during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women aged 18 to 45 years

Singleton pregnancy

Enrollment during the first trimester of pregnancy (11-13 weeks' gestation)

Ability to read and understand Turkish

Willingness to participate and provide written informed consent

Exclusion Criteria:

High-risk pregnancy, including but not limited to:

Preeclampsia

Threatened preterm labor

Placenta previa

History of pelvic surgery that may affect sexual function

Diagnosed psychiatric disorder or current use of medications that may affect sexual function/libido

Incomplete questionnaire responses at any assessment time point

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of healthy pregnant women with singleton pregnancies who are followed at a tertiary care hospital and enrolled during the first trimester of pregnancy. Participants include women who self-select to participate in instructor-led prenatal Pilates and those who do not engage in structured exercise during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) Total Score | Baseline (first trimester; 11-13 weeks' gestation), second trimester (20-24 weeks' gestation), and third trimester (32-36 weeks' gestation).
  The Female Sexual Function Index (FSFI) is a validated 19-item self-report questionnaire assessing female sexual function across six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. The FSFI total score ranges from 2.0 to 36.0, with higher scores indicating better sexual function. The FSFI total score will be collected via online questionnaires.

SECONDARY OUTCOMES:
Female Sexual Distress Scale-Revised (FSDS-R) Total Score | Baseline (first trimester; 11-13 weeks' gestation), second trimester (20-24 weeks' gestation), and third trimester (32-36 weeks' gestation).
  The Female Sexual Distress Scale-Revised (FSDS-R) is a validated 13-item self-report questionnaire designed to assess sexually related personal distress in women. The FSDS-R total score ranges from 0 to 52, with higher scores indicating greater sexual distress. The FSDS-R total score will be collected via online questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Gökçenur Karakelleoğlu, Principal Investigator — Istanbul Okan University Hospital, Department of Obstetrics and Gynecology
Locations (1):
- Istanbul Okan University Hospital, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to participant privacy concerns and the sensitive nature of questionnaire-based sexual health information.

DOCUMENTS (1):
  • Informed Consent Form: Informed Consent Form (Version 1.0 - 04 Feb 2026) (2026-02-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT07403994/ICF_000.pdf